CLINICAL TRIAL: NCT05468138
Title: PD-1 Antibody Adjuvant Therapy for Patients With MSI-H Advanced Gastric or Gastroesophageal Junction Cancer After Radical Surgery With D2 Dissection: a Phase II Single-center, Three-arm, Randomized Controlled Clinical Trial
Brief Title: PD-1 Antibody Adjuvant Therapy for GC Patients With MSI-H After D2 Radical Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Dazhi Xu, the chief of department of gastric surgery at Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAMHG
Record Dates: First submitted 2022-07-16; First posted 2022-07-21 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: MSI-H; PD-1 Immunotherapy; Gastric Cancer; Adjuvant Therapy
Keywords: gastric cancer; MSI-H; PD-1 Immunotherapy; adjuvant therapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — XELOX; Observation; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adjuvant chemotherapy(SOX or XELOX ) (Active Comparator): 8 cycles of adjuvant SOX or XELOX should be performed within 8 weeks after receiving standard gastrectomy with D2 lymphadenectomy.
  SOX: S-1：40~60mg bid，d1~14 q3W oxaliplatin：130mg/m2，iv drip for 2h，d1,q3W 8 cycles (6 months) XELOX: capecitabine：1000 mg/m2 ，bid, d1~14 q3W oxaliplatin：130mg/m2，iv drip for 2h，d1,q3W 8 cycles (6 months)
  Interventions: Drug: SOX; Drug: XELOX
- Observation (Experimental): After receiving standard gastrectomy with D2 lymphadenectomy, regular follow-up every 3 months alone. Abdomen/chest CT scan will be performed every 6 months after surgery.
  Interventions: Other: Observation
- PD-1 immunotherapy (Experimental): Adjuvant treatment with PD-1 antibody every 3 weeks(maximum 1 years) should be performed within 8 weeks after receiving standard gastrectomy with D2 lymphadenectomy.
  PD-1 antibody: Sintilimab at a dose of 200 mg every 3 weeks for 16 cycles or Nivolumab at a dose of 360 mg every 3 weeks for 16 cycles
  Interventions: Drug: PD-1 antibody

INTERVENTIONS:
Drug: SOX — Drug: Tegafur-Gimeracil-Oteracil Potassium The dose of S-1 is according to body-surface area (BSA): patients with a BSA of less than 1.25 m2 received 80 mg daily; those with a BSA of 1.25 m2 or more but less than 1.5 m2 received 100 mg daily; and those with a BSA of 1.5 m2 or more received 120 mg daily. oxaliplatin 130mg/m2, intravenously, on day 1.
  Drug: Oxaliplatin The dose of oxaliplatin is according to body-surface area (BSA): 130mg/m2, intravenously, on day 1.
  Arms: Adjuvant chemotherapy(SOX or XELOX )
Drug: XELOX — Drug: Capecitabine 1000mg/m2, orally, twice per day, from day 1 to day 14, Q3W. Drug: Oxaliplatin The dose of oxaliplatin is according to body-surface area (BSA): 130mg/m2, intravenously, on day 1.
  Arms: Adjuvant chemotherapy(SOX or XELOX )
Other: Observation — follow up and Observation alone. Abdomen/chest CT scan will be performed every 6 months after surgery.
  Arms: Observation
Drug: PD-1 antibody — Sintilimab at a dose of 200 mg every 3 weeks for 16 cycles or Nivolumab at a dose of 360 mg every 3 weeks for 16 cycles
  Arms: PD-1 immunotherapy

SUMMARY:
Approximately 5% to 10% of gastric cancers have MSI-H/dMMR. According to the results of retrospective analysis of CLASSIC and MAGIC, MSI-H/dMMR was a good prognosis and potential negative predictor of adjuvant chemotherapy for resectable gastric cancer. GC patients with MSI-H/dMMR were relatively insensitive to chemotherapy. The prognosis of these patients receiving routine postoperative adjuvant chemotherapy was worse than that with surgery alone. However, these patients were sensitive to immunotherapy. MSI-H/dMMR is one of the most important biomarkers to predict the efficacy of immunotherapy for GC. In this study, patients with MSI-H locally advanced gastric adenocarcinoma after radical surgery with D2 dissection would be randomly treated with conventional adjuvant chemotherapy, PD-1 monoclonal antibody immunotherapy or follow-up observation. We intend to demonstrate that the prognosis of MSI-H GC patients after D2 radical gastrectomy receiving PD-1 monoclonal antibody immunotherapy would be better than that with standard postoperative adjuvant chemotherapy and follow-up observation.

DETAILED DESCRIPTION:
We intend to demonstrate that the prognosis of MSI-H GC patients after D2 radical gastrectomy receiving PD-1 monoclonal antibody immunotherapy would be better than that with standard postoperative adjuvant chemotherapy and follow-up observation.

ELIGIBILITY:
Inclusion Criteria:

1. Written (signed) informed consent;
2. D2 radical gastrectomy for gastric cancer
3. Postoperative pathology confirmed II-IIIc stage gastric adenocarcinoma with dMMR/MSI-H status;
4. Female or male, 18-75 years;
5. ECOG 0-1, no surgery contraindications;
6. No initial treatment (radiotherapy / chemotherapy / immunotherapy).;
7. Esophagus not involved ≥ 3cm;
8. Basic diseases without thyroid and cardiopulmonary dysfunction
9. Adequate hematological, liver, renal and coagulation function; 1) Platelet (PLT) count ≥100,000 /mm3; 2) Neutrophil count (ANC) ≥1,500 /mm3; 3) Hemoglobin (Hb) level ≥9.0 g/dl; 4) International normalized ratio (INR) ≤1.5; 5) Prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤1.5×ULN; 6) Glycosylated hemoglobin (HbA1c) <7.5%; 7) Total bilirubin (TBIL) level ≤1.5×ULN; 8) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) level ≤2.5×ULN (≤5×ULN in case of liver metastasis); 9) Alkaline phosphatase level ≤2.5×ULN (≤5×ULN in case of liver metastasis); 10) Serum creatinine (Cr) level ≤1.5×ULN and creatinine clearance ≥60 ml/min; 11) Thyroid stimulating hormone (TSH) ≤ULN; 12) Normal serum free thyroid hormone (T4); 13) Normal serum free triiodothyronine (T3); 14) Serum amylase ≤1.5×ULN; 15) Lipase ≤1.5×ULN.
10. Females of child bearing age must have a negative pregnancy test, and have to take contraception measures and avoid breast feeding during the study and for 3 months after the last dose; male subjects must agree to taken contraception measures during the study and for 3 months after the last dose.

Exclusion Criteria:

1. Known allergy to study drug or excipients, or allergy to similar drugs;
2. Patients with active malignant tumor in recent 2 years, except the tumor studied in this research or cured localized tumor like resected basal cell or squamous cell skin cancer, superficial bladder cancer, cervical or breast carcinoma in situ;
3. Uncontrollable pleural effusion, pericardial effusion, or ascites in 2 weeks before recruitment;
4. The patient has a serious history of heart disease, including congestive heart failure, uncontrollable arrhythmia, unstable angina pectoris, myocardial infarction, severe heart valve disease and intractable hypertension;
5. Unable to swallow study drug;
6. Prior chemotherapy, radiotherapy for gastric cancer;
7. Prior therapy with a PD-1, anti-PD-Ligand 1 (PD-L1) or CTLA-4 agent;
8. Prior therapy with tyrosine kinase inhibitor within 2 weeks.
9. Concurrent medical condition requiring the use of cortisol (>10mg/day Prednisone or equivalent dose) or other systematic immunosuppressive medications within 14 days before the study treatment. Except: inhalation or topical corticosteroids. Doses > 10 mg/day prednisone or equivalent for replacement therapy;
10. Have vaccination with attenuated live vaccines within 4 weeks prior to initiation of the study treatment or plan to vaccinate during the study;
11. Poorly controlled hypertension or diabetes;
12. With bleeding tendency, or evident hemoptysis or other hemorrhagic events (e.g. gastrointestinal hemorrhage, hemorrhagic gastric ulcer) within 2 months prior to initiation of study treatment, or presence of hereditary or acquired bleeding or thrombotic tendency (e.g. hemophilia, coagulopathy, thrombocytopenia, etc.), or current/long-term thrombolytic or anticoagulant therapy (except aspirin ≤100 mg/day);
13. Present or history of any autoimmune disease;
14. With active tuberculosis or receiving previous anti-tuberculosis therapy within one year;
15. Diagnosed with interstitial pneumonia, non-infectious pneumonia, pulmonary fibrosis, acute lung disease;
16. Pregnancy or breast feeding;
17. Human immunodeficiency virus (HIV) infection (HIV antibody positive), or active hepatitis C virus (HCV) infection (HCV antibody positive), or active hepatitis B virus (HBV) infection (HBsAg or HBcAb positive, and HBV-DNA ≥2000 IU/ml (copies/ml)), or other severe infection requiring systemic antibiotic treatment, or unexplained body temperature >38.5℃ during screening period/before study treatment;
18. Patients with other severe acute or chronic conditions that may increase the risk of participation in the study and study treatment, or may interfere with interpretation of study results, and judged by the investigator as not suitable for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2022-08-25 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
3 year Disease Free Survival | 3 years
  3-year DFS

SECONDARY OUTCOMES:
morbidity | 1 year
  safety of PD1 antibody therapy
mortality | 1 year
  safety of PD1 antibody therapy
adverse events during PD1 therapy | 1 year
  safety of PD1 antibody therapy
5 year Overall Survival | 5 years
  5-year OS

CONTACTS AND LOCATIONS:
Locations (1):
- Dazhi Xu, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pietrantonio F, Miceli R, Raimondi A, Kim YW, Kang WK, Langley RE, Choi YY, Kim KM, Nankivell MG, Morano F, Wotherspoon A, Valeri N, Kook MC, An JY, Grabsch HI, Fuca G, Noh SH, Sohn TS, Kim S, Di Bartolomeo M, Cunningham D, Lee J, Cheong JH, Smyth EC. Individual Patient Data Meta-Analysis of the Value of Microsatellite Instability As a Biomarker in Gastric Cancer. J Clin Oncol. 2019 Dec 10;37(35):3392-3400. doi: 10.1200/JCO.19.01124. Epub 2019 Sep 12. PMID 31513484
- [Result] Choi YY, Kim H, Shin SJ, Kim HY, Lee J, Yang HK, Kim WH, Kim YW, Kook MC, Park YK, Kim HH, Lee HS, Lee KH, Gu MJ, Choi SH, Hong S, Kim JW, Hyung WJ, Noh SH, Cheong JH. Microsatellite Instability and Programmed Cell Death-Ligand 1 Expression in Stage II/III Gastric Cancer: Post Hoc Analysis of the CLASSIC Randomized Controlled study. Ann Surg. 2019 Aug;270(2):309-316. doi: 10.1097/SLA.0000000000002803. PMID 29727332
- [Result] Smyth EC, Wotherspoon A, Peckitt C, Gonzalez D, Hulkki-Wilson S, Eltahir Z, Fassan M, Rugge M, Valeri N, Okines A, Hewish M, Allum W, Stenning S, Nankivell M, Langley R, Cunningham D. Mismatch Repair Deficiency, Microsatellite Instability, and Survival: An Exploratory Analysis of the Medical Research Council Adjuvant Gastric Infusional Chemotherapy (MAGIC) Trial. JAMA Oncol. 2017 Sep 1;3(9):1197-1203. doi: 10.1001/jamaoncol.2016.6762. PMID 28241187
- [Result] Le DT, Uram JN, Wang H, Bartlett BR, Kemberling H, Eyring AD, Skora AD, Luber BS, Azad NS, Laheru D, Biedrzycki B, Donehower RC, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Duffy SM, Goldberg RM, de la Chapelle A, Koshiji M, Bhaijee F, Huebner T, Hruban RH, Wood LD, Cuka N, Pardoll DM, Papadopoulos N, Kinzler KW, Zhou S, Cornish TC, Taube JM, Anders RA, Eshleman JR, Vogelstein B, Diaz LA Jr. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20. doi: 10.1056/NEJMoa1500596. Epub 2015 May 30. PMID 26028255
- [Result] Chalabi M, Fanchi LF, Dijkstra KK, Van den Berg JG, Aalbers AG, Sikorska K, Lopez-Yurda M, Grootscholten C, Beets GL, Snaebjornsson P, Maas M, Mertz M, Veninga V, Bounova G, Broeks A, Beets-Tan RG, de Wijkerslooth TR, van Lent AU, Marsman HA, Nuijten E, Kok NF, Kuiper M, Verbeek WH, Kok M, Van Leerdam ME, Schumacher TN, Voest EE, Haanen JB. Neoadjuvant immunotherapy leads to pathological responses in MMR-proficient and MMR-deficient early-stage colon cancers. Nat Med. 2020 Apr;26(4):566-576. doi: 10.1038/s41591-020-0805-8. Epub 2020 Apr 6. PMID 32251400